CLINICAL TRIAL: NCT04395755
Title: Impact of COVID-19 Pandemic on the Psychological Status of Infertile Patients Who Had in Vitro Fertilization Treatment Interrupted or Postponed
Brief Title: Impact of COVID-19 on Psychological Status in Case of IVF Interrupted or Postponed
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Principal investigator, Ospedale Policlinico San Martino
Other Study IDs: COVID-19-NOIVF
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Infertility, Female; ART; IVF; COVID-19
MeSH Terms: conditions — Infertility, Female; COVID-19 | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile women who had the IVF treatment postponed or delayed
  Interventions: Behavioral: Generalized Anxiety Disorder-7 (GAD-7); Behavioral: Patient Health Questionnaire-9 (PHQ-9)

INTERVENTIONS:
Behavioral: Generalized Anxiety Disorder-7 (GAD-7) — The GAD-7 is useful in primary care and mental health settings as a screening tool and symptom severity measure for the four most common anxiety disorders.
Behavioral: Patient Health Questionnaire-9 (PHQ-9) — The PHQ-9 is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.

SUMMARY:
Infertility is a severely distressing experience for many couples. Depression and anxiety are psychological disorders associated with infertility, and they may worsen during infertility treatments.

This study times to understand the changes in the psychological status of infertile patients who had in vitro fertilization (IVF) treatment interrupted or postponed because of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* patients with IVF treatment interrupted or delayed during COVID-19 pandemic
* patients with signed informed consent
* patients with more than 18 years

Exclusion Criteria:

* patients with already diagnosed psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IVF treatment interrupted or delayed during COVID-19 pandemic
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Severity of anxiety | 1-4 weeks after communication of interrupted or delayed IVF
Severity of depression | 1-4 weeks after communication of interrupted or delayed IVF

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alviggi C, Esteves SC, Orvieto R, Conforti A, La Marca A, Fischer R, Andersen CY, Buhler K, Sunkara SK, Polyzos NP, Strina I, Carbone L, Bento FC, Galliano D, Yarali H, Vuong LN, Grynberg M, Drakopoulos P, Xavier P, Llacer J, Neuspiller F, Horton M, Roque M, Papanikolaou E, Banker M, Dahan MH, Foong S, Tournaye H, Blockeel C, Vaiarelli A, Humaidan P, Ubaldi FM; POSEIDON (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number) group. COVID-19 and assisted reproductive technology services: repercussions for patients and proposal for individualized clinical management. Reprod Biol Endocrinol. 2020 May 13;18(1):45. doi: 10.1186/s12958-020-00605-z. PMID 32404170
- [Derived] Barra F, La Rosa VL, Vitale SG, Commodari E, Altieri M, Scala C, Ferrero S. Psychological status of infertile patients who had in vitro fertilization treatment interrupted or postponed due to COVID-19 pandemic: a cross-sectional study. J Psychosom Obstet Gynaecol. 2022 Jun;43(2):145-152. doi: 10.1080/0167482X.2020.1853095. Epub 2020 Nov 30. PMID 33252292